CLINICAL TRIAL: NCT00151164
Title: Thymic Tolerance in Pediatric Heart Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to failure to control sufficient patients in the active arm, this study has now been closed.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double
Other Study IDs: 551; P50HL074732-04 (NIH); 0404019
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2008-01

CONDITIONS: Heart Transplantation
Keywords: transplantation tolerance; thymus; bone marrow; pediatric heart transplantation

INTERVENTIONS:
Procedure: donor bone marrow cell injection into thymus gland

SUMMARY:
The investigators hypothesize that injecting donor bone marrow cells into the recipient thymus gland at the time of heart transplantation in children will prove to be feasible and safe. They further hypothesize that recipients receiving donor bone marrow will experience less acute rejection events with reduced long-term requirements for immunosuppressive medications when compared to controls who do not receive marrow but who are managed under an identical immunosuppressive protocol.

ELIGIBILITY:
Inclusion Criteria:

* Less than 21 years of age at listing
* Listed for primary orthotopic heart transplant at Children's Hospital of Pittsburgh, between 04/01/04 and 03/31/08

Exclusion Criteria:

* History of prior transplant
* Listed for multi-organ transplant
* Sensitized against human HLA tissue types
* Documentation of total thymomectomy during a prior surgery

Ages: 1 Day to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2004-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Determine if intra-thymic inoculation of donor bone marrow cells at time of heart transplantation in children will reduce frequency of acute rejection as well as long-term requirements of immunosuppressive medications when compared to control patients

SECONDARY OUTCOMES:
Compare results of serial in vitro immunological monitoring among patients receiving intra-thymic bone marrow and controls

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Webber, MBChB, Principal Investigator — University of Pittsburgh Medical School
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States